CLINICAL TRIAL: NCT01008709
Title: Minimally Invasive Urologic Surgery Clip Evaluation: Can We Improve Our Surgical Technique, Reduce Costs and Waste With the Aesculap U-clip Versus the Tele-Flex Hemolock Clip?
Brief Title: Comparison Study of Two Different Surgical Clips During Laparoscopic Urologic Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Stanley Duke Herrell, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 090917
Record Dates: First submitted 2009-10-30; First posted 2009-11-06 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Prostatectomy; Nephrectomy; Laparoscopy; Robotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Teleflex HemoLock clip (Placebo Comparator): Patients randomized to the Aesculap U-clip device or the HemoLock clip will undergo their respective surgery (robotic prostatectomy and laparoscopic and robotic renal surgery) as per standard protocols. During the surgical procedure, when primary vascular control is warranted the appropriate clip to which the patient has been randomized will be utilized. Immediate assessment of the vascular pedicle will subsequently occur
  Interventions: Device: Teleflex HemoLock clip
- Aesculap U-Clip (Active Comparator): Patients randomized to the Aesculap U-clip device or the HemoLock clip will undergo their respective surgery (robotic prostatectomy and laparoscopic and robotic renal surgery) as per standard protocols. During the surgical procedure, when primary vascular control is warranted the appropriate clip to which the patient has been randomized will be utilized. Immediate assessment of the vascular pedicle will subsequently occur.
  Interventions: Device: Aesculap U-clip

INTERVENTIONS:
Device: Teleflex HemoLock clip — Patients randomized to the Aesculap U-clip device or the HemoLock clip will undergo their respective surgery (robotic prostatectomy and laparoscopic and robotic renal surgery) as per standard protocols. During the surgical procedure, when primary vascular control is warranted the appropriate clip to which the patient has been randomized will be utilized. Immediate assessment of the vascular pedicle will subsequently occur; if hemostasis is not adequate, additional clipping, endomechanical stapling or suture ligation will then be performed as necessary.
  Arms: Teleflex HemoLock clip
Device: Aesculap U-clip — Patients randomized to the Aesculap U-clip device or the HemoLock clip will undergo their respective surgery (robotic prostatectomy and laparoscopic and robotic renal surgery) as per standard protocols. During the surgical procedure, when primary vascular control is warranted the appropriate clip to which the patient has been randomized will be utilized. Immediate assessment of the vascular pedicle will subsequently occur; if hemostasis is not adequate, additional clipping, endomechanical stapling or suture ligation will then be performed as necessary.
  Arms: Aesculap U-Clip

SUMMARY:
Intracorporeal suturing and knot tying during robotic prostatectomy and laparoscopic and robotic renal surgery have historically been considered the most technically challenging and time consuming aspects of these procedures. With improved operative technique as well as the use of innovative surgical devices, vascular control during these surgeries is often less cumbersome as compared with traditional techniques. Current standard methods of hemostasis include the use of clips, of which the most popular design is the Hemolock, a locking, nonabsorbable plastic clip, or the use of the very expensive endomechanical stapler. Unfortunately while they are associated with time savings in the operating room, there is a great deal of disposable costs associated with these various devices as well as a not insignificant device malfunction rate reported in the literature. The aim of this case-controlled study is to evaluate the Aesculap U-clip device compared to our current technique of vascular control using the Teleflex Hemolock clip device during minimally invasive genitourinary surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years old with genitourinary malignancy either prostate cancer or kidney renal masses undergoing minimally invasive genitourinary organ removal will be included in this small pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
significant difference in clip misfire and misapplication rates | 1month

SECONDARY OUTCOMES:
blood loss / need for transfusion | 1 month
OR time | 1 day
Need for repeat procedure | 1 month
number of clips used | 1 day
surgeon impression of the ease of application | 1 day
predicted cost differential (or at least charge differential) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: S. Duke Herrell, MD, Principal Investigator — Vanderbilt University Department of Urologic Surgery
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Meng MV. Reported failures of the polymer self-locking (Hem-o-lok) clip: review of data from the Food and Drug Administration. J Endourol. 2006 Dec;20(12):1054-7. doi: 10.1089/end.2006.20.1054. PMID 17206901
- [Background] Hsi RS, Saint-Elie DT, Zimmerman GJ, Baldwin DD. Mechanisms of hemostatic failure during laparoscopic nephrectomy: review of Food and Drug Administration database. Urology. 2007 Nov;70(5):888-92. doi: 10.1016/j.urology.2007.06.1116. Epub 2007 Oct 24. PMID 17919695